CLINICAL TRIAL: NCT02551679
Title: A Randomized Double Blind Placebo Controlled Clinical Study to Assess Blood-Derived Autologous Angiogenic Cell Precursor Therapy in Patients With Critical Limb Ischemia (ACP-CLI)
Brief Title: ACP-01 in Patients With Critical Limb Ischemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hemostemix (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HS 12-01.; NCT02140931 (obsolete NCT alias)
Record Dates: First submitted 2015-09-14; First posted 2015-09-16 (Estimated); Results first posted 2023-11-18 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Critical Limb Ischemia
Keywords: Stem cells; Autologous; Vascular disease; Peripheral arterial disease; Regenerative medicine; Amputation
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia; Vascular Diseases; Peripheral Arterial Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ACP-01 (Active Comparator): Injection into lower extremity
  Interventions: Biological: ACP-01
- Placebo (Placebo Comparator): Injection into lower extremity
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: ACP-01 — Injection into lower extremity
  Arms: ACP-01
Biological: Placebo — Injection into lower extremity
  Arms: Placebo

SUMMARY:
The primary objective of this study is to determine the efficacy and safety of intramuscular injection of ACP-01, comprised of blood-derived autologous ACPs, in subjects with critical limb ischemia who are receiving standard of care therapy and have no endovascular or surgical revascularization options.

DETAILED DESCRIPTION:
This prospective, randomized, double-blind, placebo controlled study will assess the efficacy and safety of autologous ACPs administered intramuscularly into the lower extremity of subjects with CLI who lack surgical or endovascular revascularization options.

A total of approximately 95 subjects will be randomized to treatment with ACP-01 or placebo using a 2:1 randomization scheme, respectively, stratified by site.

The study will continue until all subjects treated experience the study event (either de novo gangrene, doubling of wound size, major amputation, or death) or are event-free for at least 26 weeks. Subjects treated will be followed for no longer than 52 weeks.

One futility analysis for potentially stopping study enrollment will be performed.

Subjects treated at each investigative site will provide written informed consent prior to the conduct of any study-related procedures. Thereafter, they will be screened and those meeting the inclusion/exclusion criteria will be enrolled into the trial and undergo all the study procedures including intramuscular injection of the investigational medicinal product (IMP = ACP-01 or placebo). The IMP will be administered in addition to any conventional treatment the subject is receiving.

The control group will receive placebo injections into the lower extremity to ensure blinding of the assessors and the subjects.

The placebo will consist of the same medium used in the ACP product suspension.

The study consists of four periods: Screening period, Treatment period, Acute safety follow-up and Long term follow-up periods. The total duration of study participation, including follow-up, is at least 26 weeks. Subjects will be followed for up to 52 weeks and at least until the last subject has completed his/her 26 week visit.

ELIGIBILITY:
Inclusion Criteria:

* Subject is diagnosed with critical limb ischemia.
* Subject has hemodynamic indicators of severe peripheral arterial occlusive disease.
* Subject is not a candidate for standard revascularization treatment options for peripheral arterial disease.
* Subject must be on standard of care medical therapy for peripheral vascular disease.
* Male or female age 18 and above.
* Non-pregnant, non-lactating female.
* Subject is able to understand and provide voluntary signed informed consent.

Exclusion Criteria:

* Uncorrected aorto-iliac occlusive disease.
* Subjects who, in the opinion of the investigator, have a vascular disease prognosis that indicates they would require a major amputation in a time frame shortly after administration of the IMP (investigational drug or placebo).
* Advanced Critical Limb Ischemia (CLI) presenting as severe ischemic or dry gangrene.
* Lower extremity non-treated active infection.
* Hypercoagulable state.
* Subject received a blood transfusion during the previous 4 weeks (to exclude the potential of non-autologous ACPs in the harvested blood).
* Inability to communicate that may interfere with clinical evaluation.
* Recent major non-vascular operation.
* Myocardial infarction or uncontrolled myocardial ischemia or persistent severe heart failure.
* Severe aortic stenosis.
* Renal failure.
* Hepatic failure.
* Anemia.
* Major stroke.
* Diagnosis of malignancy.
* Concurrent chronic or acute infectious disease and uncontrolled infectious symptoms.
* Severe concurrent disease (other than Peripheral Vascular Disease (PAD)).
* Bleeding diathesis.
* Participation at the same time in another investigational product or device study.
* Chronic cytotoxic drug treatment.
* Life expectancy of less than 6 months.
* Subject unlikely to be available for follow-up.
* Acute worsening of CLI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2020-04 (Actual); Study Completion 2021-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (19):
- United States (16):
  - UC Davis CTSC Clinical Research Center, Sacramento, California
  - Rocky Mountain Regional VA Medical Center, Aurora, Colorado
  - University of Florida, Gainesville, Florida
  - Clinovation Research, LLC, Miami, Florida
  - Clinical Research of Central Florida, Winter Haven, Florida
  - Decatur Memorial Hospital, Decatur, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Moses H. Cone Memorial Hospital, Greensboro, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Temple University Hosptial, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Houston Methodist DeBakey Heart & Vascular Center, Houston, Texas
  - Clinical Trials of Texas, Inc. (CTT), San Antonio, Texas
- Canada (3):
  - Vancouver General Hospital, Vancouver, British Columbia
  - London Health Sciences Centre, London, Ontario
  - Toronto General Hospital, Toronto, Ontario

REFERENCES:
- See also: Hemostemix Inc. website — http://www.hemostemix.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ACP-01 | Placebo
Started | 46 | 21
Completed | 27 | 19
Not Completed | 19 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ACP-01 | Placebo | Total
Number analyzed (Participants) | 46 | 21 | 67
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 4 | 14
  >=65 years | 36 | 17 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 70 (13.19) | 72 (9.86) | 70.9 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 8 | 25
  Male | 29 | 13 | 42
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 43 | 18 | 61
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 8 | 5 | 13
  United States | 38 | 16 | 54

OUTCOME MEASURES:

1. Primary Outcome: Wound Size, Amputation or Survival
Description: Number of subject with doubling of wound size, major amputation or death
Time Frame: Baseline vs. 1 year
Population: The primary endpoint was time from treatment to either de-novo gangrene in the treated limb, or doubling of wound size in the treated limb, or major amputation in the treated limb, or death.
Measure: Number; unit: participants
Groups:
- ACP-01: Injection into lower extremity
  ACP-01: Injection into lower extremity
  The primary endpoint was time from treatment to either de-novo gangrene in the treated limb, or doubling of wound size in the treated limb, or major amputation in the treated limb, or death. The primary outcome was analyzed using a Cox proportional hazards model to generate an HR adjusted for recruitment site. Kaplan-Meier survival curves were created for visual presentation of time-to-event comparisons. For subjects who were lost to follow-up or completed 12 months study visit without a study event, the time to event was censored by the subject's last follow-up date in the study.
- Placebo: Injection into lower extremity
  Placebo: Injection into lower extremity
  The primary endpoint was time from treatment to either de-novo gangrene in the treated limb, or doubling of wound size in the treated limb, or major amputation in the treated limb, or death. The primary outcome was analyzed using a Cox proportional hazards model to generate an HR adjusted for recruitment site. Kaplan-Meier survival curves were created for visual presentation of time-to-event comparisons. For subjects who were lost to follow-up or completed 12 months study visit without a study event, the time to event was censored by the subject's last follow-up date in the study.
Arm/Group | ACP-01 | Placebo
Number analyzed (Participants) | 46 | 21
participants | 12 | 3
Statistical Analysis 1: Comparison: ACP-01 vs Placebo; The primary hypothesis of this study is that ACP-01 is superior to placebo in terms of the earlier time from treatment with Investigational Medicinal Product (IMP) to either de-novo gangrene, or doubling of wound size, or major amputation, or death; Test type: Superiority; p = 0.258, ANCOVA; Cox Proportional Hazard = 2.046, 95% CI 2-sided [0.577 to 7.255]

2. Secondary Outcome: Pain Level
Description: Change in pain score according to the Visual Analog Scale (VAS) for Pain. The visual VAS is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between the two ends of the scale-"no pain" on the left end (0 cm) of the scale and the "worst pain" on the right end of the scale (10 cm). Measurements from the starting point (left end) of the scale to the subjects' marks are recorded in centimeters and are interpreted as their pain. The values ar used to track pain progression for a subject and to compare pain between subjects.
Time Frame: Baseline vs. 1 year
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | ACP-01 | Placebo
Number analyzed (Participants) | 46 | 21
units on a scale | 38.75 (9.479) | 44.44 (14.036)

3. Secondary Outcome: Ulcer Size
Description: Change in ulcer size
Time Frame: Baseline vs. 1 year
Measure: Least Squares Mean (Standard Error); unit: cm^2
Arm/Group | ACP-01 | Placebo
Number analyzed (Participants) | 46 | 21
cm^2 | 1.6 (1.07) | 1.8 (0.59)

4. Other Pre Specified Outcome: Change From Baseline in the Dose and Quantity of Analgesic Drugs Used by the Subject
Time Frame: 1 - 52 wks
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Reduction in Total Hospitalization Time of Subjects Treated With ACP-01 Compared to Subjects Treated With Placebo
Time Frame: 1 - 52 wks
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Change From Baseline in Quality of Life
Description: Change in quality of life according to the Vascular Quality of Life Questionnaire.
Time Frame: 1 - 52 wks
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Change From Baseline in Ankle Pressure
Time Frame: 1 - 52 wks
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Change From Baseline in Toe Pressure
Time Frame: 1 - 52 wks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | ACP-01 | Placebo
All-Cause Mortality (participants affected / at risk) | 5/46 | 1/21
Serious Adverse Events (participants affected / at risk) | 2/46 | 1/21
Other Adverse Events (participants affected / at risk) | 0/46 | 0/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ACP-01 (N=46) | Placebo (N=21)
acute myocardial infarction (Cardiac disorders) | 2 (2) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Cardiovascular disorder (Cardiac disorders) | 1 (1) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Gangrene (Infections and infestations) | 2 (2) | 1 (1)
Localized infection (Infections and infestations) | 1 (1) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Vascular stent infection (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2019-10-18): https://cdn.clinicaltrials.gov/large-docs/79/NCT02551679/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-01): https://cdn.clinicaltrials.gov/large-docs/79/NCT02551679/SAP_001.pdf